CLINICAL TRIAL: NCT01213368
Title: Double Blind, Randomized, Placebo Controlled Dose Ranging Study of the Efficacy and Safety of Dronedarone (SR33589B) at 300, 400, or 600 mg BID for the Control of Ventricular Rate in Japanese Patients With Permanent Atrial Fibrillation
Brief Title: Dose Ranging Study of Dronedarone for the Control of Ventricular Rate in Japanese Patients With Permanent Atrial Fibrillation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRI10939; U1111-1116-9409 (Other: (UTN))
Record Dates: First submitted 2010-09-30; First posted 2010-10-04 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dronedarone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- dronedarone 300 mg (Experimental): Dronedarone, 100mg + 200mg tablets twice daily, administered with food.
  Interventions: Drug: DRONEDARONE (SR33589)
- dronedarone 400 mg (Experimental): Dronedarone, 400mg tablets twice daily, administered with food.
  Interventions: Drug: DRONEDARONE (SR33589)
- dronedarone 600 mg (Experimental): Dronedarone, 400mg + 200mg tablets twice daily, administered with food.
  Interventions: Drug: DRONEDARONE (SR33589)
- placebo (Placebo Comparator): Matching placebo tablets twice daily, administered with food.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: DRONEDARONE (SR33589) — Pharmaceutical form: tablets
  Route of administration: oral
  Arms: dronedarone 300 mg; dronedarone 400 mg; dronedarone 600 mg
Drug: placebo — Pharmaceutical form: tablets
  Route of administration: oral
  Arms: placebo

SUMMARY:
Primary Objective:

- To assess the efficacy of dronedarone versus placebo for the control of ventricular rate in patients with permanent Atrial Fibrillation (AF).

Secondary Objective:

* To assess the safety and tolerability of dronedarone after repeated oral doses of 300 mg, 400 mg, or 600 mg twice daily in the selected population.
* To document SR33589 and SR35021 trough plasma levels at steady state.

DETAILED DESCRIPTION:
The study period per patient is approximatively 1 month broken down as follows:

* Screening period up to 7 days,
* Treatment period of 14 days,
* Follow-up period of 10 days.

ELIGIBILITY:
Inclusion criteria:

* Patients of aged 20 years or more.
* Permanent Atrial Fibrillation [AF] (defined as duration of AF > 6 months) for which cardioversion is not considered and with resting ventricular heart rate ≥ 80 bpm at screening.

Exclusion criteria:

* Unstable angina pectoris.
* History of torsades de pointes.
* Prolonged QT corrected interval (≥ 500 ms).
* Third degree atrioventricular block (AVB) on the screening ECG while in AF or, documentation on previous ECGs while in sinus rhythm of PR-interval > 0.28 sec or high degree AVB (2nd degree or higher) or, significant sinus node disease (documented pause ≥ 3 sec) - without a permanent pacemaker implanted.
* Congestive Heart Failure (CHF) of New York Heart Association classification (NYHA) class IV or recent (within 1 month prior to randomization) unstable NYHA class III.
* Treatment with other class I or III anti-arrhythmic drugs.
* Patients treated with amiodarone during the 4 weeks preceding randomization.
* Clinically relevant haematologic, hepatic, gastro-intestinal, renal, pulmonary, endocrinologic (in particular thyroid) or psychiatric disease.
* Hypokalemia and hypomagnesemia must be corrected before randomization.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2010-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean ventricular rate measured by 24-hour Holter Electrocardiogram (ECG) | Day 14

SECONDARY OUTCOMES:
Number of patients with adverse events | up to 10 days after last drug intake
Plasma trough concentrations for SR33589 | Day 14
Plasma trough concentrations for SR35021 | Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (25):
- Japan (25):
  - Investigational Site Number 392022, Hiroshima
  - Investigational Site Number 392018, Kagoshima
  - Investigational Site Number 392005, Kasama-Shi
  - Investigational Site Number 392014, Kawanishi-Shi
  - Investigational Site Number 392008, Kawasaki-Shi
  - Investigational Site Number 392007, Kisarazu-Shi
  - Investigational Site Number 392012, Kobe
  - Investigational Site Number 392013, Kobe
  - Investigational Site Number 392003, Koriyama-Shi
  - Investigational Site Number 392017, Kurume-Shi
  - Investigational Site Number 392023, Miyazaki
  - Investigational Site Number 392009, Nagano
  - Investigational Site Number 392019, Nagasaki
  - Investigational Site Number 392010, Osaka
  - Investigational Site Number 392021, Sapporo
  - Investigational Site Number 392025, Sapporo
  - Investigational Site Number 392002, Sendai
  - Investigational Site Number 392004, Shirakawa-Shi
  - Investigational Site Number 392016, Shunan-Shi
  - Investigational Site Number 392020, Suwa-Shi
  - Investigational Site Number 392006, Takasaki-Shi
  - Investigational Site Number 392001, Tomakomai-Shi
  - Investigational Site Number 392024, Toshima-Ku
  - Investigational Site Number 392015, Ube-Shi
  - Investigational Site Number 392011, Yakushi